CLINICAL TRIAL: NCT01623674
Title: Laparoscopic Skills and Cognitive Function Are Not Affected by Night Shifts in Surgeons
Status: Completed | Type: Observational
Sponsor: Herlev Hospital (Other)
Collaborators: TRYG Foundation (Other); Danish Medical Association (Other)
Responsible Party: Principal Investigator, Ilda Amirian, MD, PHD student at Unit of Surgical Gastroenterology, Herlev Hospital
Other Study IDs: Herlev-12345
Record Dates: First submitted 2012-06-18; First posted 2012-06-20 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-05

CONDITIONS: Effect of Sleep Deprivation
Keywords: Sleep deprivation in surgeons during night shifts and the effect on performance.

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urin (melatonine) Saliva (cortisol)
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study was to asses the effect of sleep deprivation during nightshift by monitoring 30 surgeons in unit of surgical gastroenterology in 4 consecutive days. The first day was pre call= day 1, second day was on call= day 2, third day was the first post call day = day 3 and fourth day was the second post call= day 4. The surgeons were monitored in order to asses how performance was on call compared to pre call and post call. The hypothesis was that they would perform worse on call than pre call, and again slightly worse post call.

DETAILED DESCRIPTION:
The surgeons wore an actigraph consecutively on all 4 days, and would fill out a sleep diary on all 4 days as well. The surgeons were heart monitored consecutively on day 1 and 2.

The surgeons were tested in a laparoscopic simulator at 8 a.m. day 1, 4 a.m. day 2, and again at 8 a.m. day 4. At the same given times they would perform the d2 test of attention and prescribe medicine in the Electronic Patient Medication system in accordance with a case they were given. Furthermore they delivered a salivary sample for the determination of salivary cortisol, at the given times.

They sampled urine from 9 pm - 9 am all 4 days, in order to measure the production of melatonin in urine.

The surgeons would fill out the Karolinska sleepiness scale, VAS (Visual Analog Scale) fatigue, VAS sleep quality and VAS general well being at 8 a.m. day 1, 4 a.m. day 2, and again at 8 a.m. day 4. The Karolinska Sleepiness scale was filled out every second hour on day 2 from 4pm - 8 am on day 3.

ELIGIBILITY:
Inclusion Criteria:

* Surgeons at surgical unit of Gastroenteroloy
* Men and women between the age of 22-50 years.

Exclusion Criteria:

* Pregnancy and breastfeeding
* Endocrine disease, medically treated
* Autoimmune disease, medically treated
* Sleep disturbance, medically treated
* Intake of alcohol within 24 hours before the study and during the entire study

Ages: 22 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Surgeons at a surgical unit of gastroenterology in Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-12; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
laparoscopic simulation | pre call and on call

SECONDARY OUTCOMES:
d2 test of attention, Karolinska Sleepiness scale, actigraphy, prescribing medication in the EPM system, HRV, urine melatonine, saliva cortisol | pre call, on call, post call, the second post call day

CONTACTS AND LOCATIONS:
Locations (1):
- University of Copenhagen, Herlev Hospital, Herlev, Herlev, Denmark

REFERENCES:
- [Derived] Amirian I, Toftegard Andersen L, Rosenberg J, Gogenur I. Decreased heart rate variability in surgeons during night shifts. Can J Surg. 2014 Oct;57(5):300-4. doi: 10.1503/cjs.028813. PMID 25265102